CLINICAL TRIAL: NCT02299336
Title: Long-Term Efficacy and Safety of Intravitreal Aflibercept Injections for the Treatment of Diabetic Macular Edema in Subjects Who Completed the Three Year VISTA-DME Trial .
Brief Title: Long-Term Efficacy & Safety of Aflibercept IVT for the Treatment of DME in Subjects Who Completed the VISTA-DME Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Greater Houston Retina Research (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Charles C Wykoff, PhD, MD, Principal Investigator, Greater Houston Retina Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The Endurance 1 Trial
Record Dates: First submitted 2014-10-15; First posted 2014-11-24 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRN (pro re nata) (Other): 2 mg intravitreal aflibercept (Eylea) PRN, focal laser administered based on pre-specified criteria, 104 weeks
  Interventions: Drug: Aflibercept; Procedure: Focal Laser

INTERVENTIONS:
Drug: Aflibercept — pro re nata (PRN)
  Other Names: Eylea
Procedure: Focal Laser — Focal laser administered based on pre-specified criteria

SUMMARY:
The Endurance Trial is a phase IV open label clinical study to assess the need for ongoing intravitreal aflibercept injections after the 3-year VISTA DME (VGFT-OD-1009; NCT01363440) end-point. Subjects will be treated with intravitreal aflibercept injections pro re nata (PRN) based on the presence of CR-DME (Clinically Relevant-DME). In addition, subjects who meet re-treatment criteria will be eligible for focal laser treatment every 90 days.

DETAILED DESCRIPTION:
The investigational product is aflibercept, which will be supplied by Regeneron Pharmaceuticals, Inc. in sterile vials for intravitreal (IVT) injection. Vials must be used (defined as entered with needle) only once. All drug supplies are to be kept under recommended storage conditions.

The injection volume will be 50μL (0.05 mL) and will be administered to the subjects by IVT injection.

Throughout the trial, subjects will be treated with intravitreal aflibercept injections PRN in the presence of CR-DME; this is defined as DME that the treating investigator believes is limiting visual function.

All subjects will initially be evaluated every 4 weeks (28 days) for CR-DME and treated PRN. If CR-DME is present the subject will receive IVT aflibercept injection. If CR-DME is not present the subject will not receive an IVT aflibercept injection and will be observed.

At any point throughout the study, once a subject has been evaluated and observed (with no IVT aflibercept) for a total of 8 weeks (3 consecutive monthly visits), the interval between visits will be increased to 8 weeks.

After an additional 24 weeks (3 consecutive visits, every 8 weeks) without an IVT aflibercept injection, the interval between visits will be increased to 12 weeks.

If a subject has recurrent CR-DME they will receive an IVT aflibercept injection and the interval between visits will reduce back to 4 weeks. Subjects can again extend the interval between visits to 8 weeks once they have not received an IVT aflibercept injection for a total of 8 weeks (3 consecutive visits) as described above. Extension to 12 weeks is then performed as above.

Starting at week 52, once a subject has extended to a 12 week interval, if CR-DME is not present the subject will not receive an IVT aflibercept injection and will be extended to a 16 week interval. Once at a 16 week interval, if CR-DME is not present the subject will not receive an IVT aflibercept injection and will be extended to a 20 week interval. At any point past a 12 week interval extension, if a subject has recurrent CR-DME they will receive an IVT aflibercept injection and the interval for the next visit will be reduced at investigator discretion to be either 12 or 16 weeks. If the interval is needed to be reduced to below 12 weeks, the subject will return to a 4 or 8 week interval, at investigator discretion and return to the protocol above.

All subjects receiving PRN IVT aflibercept injections will be evaluated for focal laser treatment beginning at week 12 through the end of the study. If the subject meets any of the criteria for focal laser treatment (FLT), fluorescein angiography (FA) will be performed to guide the focal laser treatment. Focal laser treatment and focal laser re-treatment will be administered no more than once every 90 days.

When a subject receives ≥ 2 IVT aflibercept injections in ≤ 24 weeks FLT will be applied. Once the initial session of FLT is applied subjects are eligible for FLT re-treatment after 90 days, when they have received ≥ 2 IVT aflibercept injections within the prior 90 day period.

FLT will be applied to:

1. All leaking microaneurysms.
2. Grid to all areas of diffuse leakage.
3. Grid to all areas of retinal ischemia outside of the FAZ (once ischemic areas are treated once with grid FLT, these same areas should not be treated again).
4. Laser will not be applied within the capillaries of the FAZ.

FLT will not be applied if any of the following apply and are identified:

1. Significant macular ischemia involving the foveal avascular zone (once this has been determine additional fluorescein angiography for FLT planning should not be performed and subjects will not longer be eligible for rescue FLT).
2. Treatment would be too close to the foveal avascular zone.
3. Macular edema is not related to DME (eg: postoperative CME, etc).

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet the following criteria to be eligible for inclusion in the study:

  1. Enrolled and Completed VISTA DME (VGFT-OD-1009) clinical trial
  2. Willing and able to comply with clinic visits and study-related procedures
  3. Provide signed informed consent
  4. Enrollment in the trial within 12 weeks of trial activation.

Exclusion Criteria:

* A subject who meets any of the following criteria will be excluded from the study:

  1. Prior treatment with anti-VEGF therapy in the study eye within 28 days of baseline
  2. Pregnant or breast-feeding women
  3. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

     * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Wykoff, MD, Principal Investigator — Greater Houston Retina Research
Locations (3):
- United States (3):
  - Retina Consultants of Houston/The Medical Center, Houston, Texas
  - Retina Consultants of Houston/Katy office, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arevalo JF, Sanchez JG, Wu L, Maia M, Alezzandrini AA, Brito M, Bonafonte S, Lujan S, Diaz-Llopis M, Restrepo N, Rodriguez FJ, Udaondo-Mirete P; Pan-American Collaborative Retina Study Group. Primary intravitreal bevacizumab for diffuse diabetic macular edema: the Pan-American Collaborative Retina Study Group at 24 months. Ophthalmology. 2009 Aug;116(8):1488-97, 1497.e1. doi: 10.1016/j.ophtha.2009.03.016. Epub 2009 Jul 9. PMID 19545900
- [Background] Bhagat N, Grigorian RA, Tutela A, Zarbin MA. Diabetic macular edema: pathogenesis and treatment. Surv Ophthalmol. 2009 Jan-Feb;54(1):1-32. doi: 10.1016/j.survophthal.2008.10.001. PMID 19171208
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Ferrara N. VEGF: an update on biological and therapeutic aspects. Curr Opin Biotechnol. 2000 Dec;11(6):617-24. doi: 10.1016/s0958-1669(00)00153-1. PMID 11102799
- [Background] Grover D, Li TJ, Chong CC. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD005656. doi: 10.1002/14651858.CD005656.pub2. PMID 18254088
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Moss SE, Klein R, Klein BE. Ten-year incidence of visual loss in a diabetic population. Ophthalmology. 1994 Jun;101(6):1061-70. doi: 10.1016/s0161-6420(94)31217-6. PMID 8008348
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648
- [Background] Nguyen QD, Tatlipinar S, Shah SM, Haller JA, Quinlan E, Sung J, Zimmer-Galler I, Do DV, Campochiaro PA. Vascular endothelial growth factor is a critical stimulus for diabetic macular edema. Am J Ophthalmol. 2006 Dec;142(6):961-9. doi: 10.1016/j.ajo.2006.06.068. Epub 2006 Aug 2. PMID 17046701
- [Background] Saaddine JB, Honeycutt AA, Narayan KM, Zhang X, Klein R, Boyle JP. Projection of diabetic retinopathy and other major eye diseases among people with diabetes mellitus: United States, 2005-2050. Arch Ophthalmol. 2008 Dec;126(12):1740-7. doi: 10.1001/archopht.126.12.1740. PMID 19064858
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Zhang X, Saaddine JB, Chou CF, Cotch MF, Cheng YJ, Geiss LS, Gregg EW, Albright AL, Klein BE, Klein R. Prevalence of diabetic retinopathy in the United States, 2005-2008. JAMA. 2010 Aug 11;304(6):649-56. doi: 10.1001/jama.2010.1111. PMID 20699456
- [Derived] Wykoff CC, Ou WC, Khurana RN, Brown DM, Lloyd Clark W, Boyer DS; ENDURANCE Study Group. Long-term outcomes with as-needed aflibercept in diabetic macular oedema: 2-year outcomes of the ENDURANCE extension study. Br J Ophthalmol. 2018 May;102(5):631-636. doi: 10.1136/bjophthalmol-2017-310941. Epub 2017 Aug 16. PMID 28814412

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRN (Pro re Nata)
Started | 60
Completed | 46
Not Completed | 14
Not completed — Withdrawal by Subject | 11
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60
Glycated Hemoglobin [Mean (Standard Deviation); unit: Percent] | 7.5 (1.1)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 18.6 (10.6)
Early Treatment Diabetic Retinopathy Study Best-Corrected Visual Acuity [Mean (Standard Deviation); unit: letters] — Participants were challenged with reading letters on lines of an eye chart (5 letters per line) in standardized lighting conditions. Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified.
  letters | 69.6 (13.4)
Central Retinal Thickness [Mean (Standard Deviation); unit: Microns] | 290 (88.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Intravitreal Aflibercept Injections for Subjects Who Were Enrolled and Completed the 3-year VISTA DME (VGFT-OD-1009) Trial
Description: Measured by evaluating mean number of injections required for subjects who were enrolled and completed the 3-year VISTA DME (VGFT-OD-1009) trial
Time Frame: Week 104
Measure: Mean (Standard Error); unit: injections
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 46
injections | 9.5 (6.7)

2. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study Best-corrected Visual Acuity From Baseline to Week 52 and Baseline to Week 104
Description: Evaluate the mean change over time in Early Treatment Diabetic Retinopathy Study best-corrected visual acuity at week 52 from baseline and at week 104 from baseline. Participants were challenged with reading letters on lines of an eye chart (5 letters per line) in standardized lighting conditions. Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified.
Time Frame: Week 52, Week 104
Population: All participants were included in analysis. Due to participant attrition, missed visits, and variable follow-up intervals, the population analyzed at each time point is equal to or smaller than the population still enrolled at that time point.
Measure: Mean (Standard Error); unit: letters
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
letters
  52 Weeks: number analyzed (Participants) | 54
  52 Weeks | 0.61 (1.28)
  104 Weeks: number analyzed (Participants) | 46
  104 Weeks | 0.83 (1.66)

3. Secondary Outcome: Mean Number of Intravitreal Aflibercept Injections Before and After Receiving First Focal Laser Application.
Description: Measure the role of focal laser treatment (fluorescein angiography-guided, if applicable) in decreasing the treatment burden among subjects who require ongoing aflibercept treatment in the management of diabetic macular edema.
Time Frame: Before First Focal Laser Treatment (FLT) at Week 12 or later; After First FLT at up to 104 weeks
Population: Only participants who were eligible for focal laser treatment were analyzed.
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 27
Injections
  Injections Before First Focal Laser | 7.5 (3.7)
  Injections After First Focal Laser | 6.7 (4.2)

4. Secondary Outcome: Percentage of Subjects With Gain or Loss of 0 to 5 Early Treatment Diabetic Retinopathy Study Best-corrected Visual Acuity Letters From Baseline to Week 52 and Baseline to Week 104
Description: Evaluate the percentage of subjects with a gain or loss in Early Treatment Diabetic Retinopathy Study best-corrected visual acuity letters in patients treated with aflibercept from baseline to week 52 and baseline to week 104
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Participants
  Week 52: number analyzed (Participants) | 54
  Week 52 | 35
  Week 104: number analyzed (Participants) | 46
  Week 104 | 30

5. Secondary Outcome: Mean Change in Central Retinal Thickness From Baseline to Week 52 and Baseline to Week 104.
Description: Evaluate the mean change in central retinal thickness from baseline to week 52 and baseline to week 104 in patients treated with aflibercept.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Microns
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Microns
  Week 52: number analyzed (Participants) | 54
  Week 52 | -7 (8.6)
  Week 104: number analyzed (Participants) | 46
  Week 104 | 1 (11.53)

6. Secondary Outcome: Number of Subjects With no Clinically-relevant Diabetic Macular Edema (as Defined in the Protocol) on Spectral Domain Optical Coherence Tomography From Baseline to Week 52 and Baseline to Week 104.
Description: Evaluate the number of subjects with no clinically-relevant diabetic macular edema (as defined in the protocol) on spectral domain optical coherence tomography from baseline to week 52 and baseline to week 104 in patients treated with aflibercept.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Participants
  Week 52: number analyzed (Participants) | 54
  Week 52 | 39
  Week 104: number analyzed (Participants) | 46
  Week 104 | 29

7. Secondary Outcome: Number of Subjects With Stable, Worsened, or Improved Diabetic Retinopathy
Description: Number of subjects with stable, worsened, or improved diabetic retinopathy through 104 weeks.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Participants
  Week 52: number analyzed (Participants) | 54
  Week 52: Worsened Diabetic Retinopathy | 5
  Week 52: Stable Diabetic Retinopathy | 46
  Week 52: Improved Diabetic Retinopathy | 3
  Week 104: number analyzed (Participants) | 46
  Week 104: Worsened Diabetic Retinopathy | 15
  Week 104: Stable Diabetic Retinopathy | 27
  Week 104: Improved Diabetic Retinopathy | 4

8. Secondary Outcome: Number of Subjects That Receive Focal Laser Treatment.
Description: Number of subjects that receive focal laser treatment from baseline to week 52 and from baseline to week 104.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
Participants
  Week 52: number analyzed (Participants) | 54
  Week 52 | 25
  Week 104: number analyzed (Participants) | 46
  Week 104 | 27

9. Secondary Outcome: Mean Change in Early Treatment Diabetic Retinopathy Study Best-corrected Visual Acuity Before and After Focal Laser Therapy
Description: Evaluation of the effect of laser on Early Treatment Diabetic Retinopathy Study best-corrected visual acuity outcomes. Participants were challenged with reading letters on lines of an eye chart (5 letters per line) in standardized lighting conditions. Lines became smaller as participants progressed from the top to the bottom of the chart. Participants read down the chart until they reached a row where a minimum of three letters on a line could be read, and were scored by how many letters could be correctly identified.
Time Frame: 104 weeks
Population: All participants receiving laser were included in analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 27
letters
  Before First FLT: number analyzed (Participants) | 25
  Before First FLT | 0.4 (6.2)
  After First FLT | 0.3 (11.9)

10. Secondary Outcome: Mean Change in Central Retinal Thickness Before and After First Focal Laser Treatment
Description: Evaluate the mean change in central retinal thickness before and after first focal laser treatment in patients treated with pro re nata aflibercept.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: microns
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 60
microns
  Before First FLT: number analyzed (Participants) | 25
  Before First FLT | -8.5 (52.6)
  After First FLT: number analyzed (Participants) | 27
  After First FLT | -6.8 (41.6)

11. Secondary Outcome: Role of (Ultrawide-field, if Available) Fluorescein Angiography-determined Retinal Ischemia in Predicting Past and Future Anti-VEGF Treatment Burden
Description: Mean number of injections in 52 weeks and 104 weeks based on quantification of ischemic areas
Time Frame: Week 52, Week 104
Population: This analysis was never performed because we were logistically unable to collect the data.
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 0

12. Secondary Outcome: Role of (Ultrawide-field, if Available) Fluorescein Angiography-determined Retinal Ischemia in Predicting Visual Outcomes
Description: Mean change in visual acuity from baseline to week 52 and baseline to week 104 based on quantification of ischemic areas
Time Frame: Week 52, Week 104
Population: This analysis was never performed because we were logistically unable to collect the data.
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 0

13. Secondary Outcome: Role of (Ultrawide-field, if Available) Fluorescein Angiography-determined Retinal Ischemia in Predicting Anatomic Outcomes
Description: Mean change in central retinal thickness from baseline to week 52 based on quantification of ischemic areas
Time Frame: Week 52, Week 104
Population: This analysis was never performed because we were logistically unable to collect the data.
Arm/Group | PRN (Pro re Nata)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 104 weeks.
Description: Adverse events were assessed at every study visit during the 2-year study.
Arm/Group | PRN (Pro re Nata)
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 19/60
Other Adverse Events (participants affected / at risk) | 26/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRN (Pro re Nata) (N=60)
Myocardial Infarction (Cardiac disorders) | 2 — Resulted in death of a subject.
Deep vein thrombosis (Vascular disorders) | 1
Stroke (Vascular disorders) | 2
Worsening congestive heart failure (Cardiac disorders) | 1
Acute vision loss secondary to vitreous hemorrhage (Eye disorders) | 2
Acute vision loss due to worsening cataract (Eye disorders) | 1
Worsening staph infection (Infections and infestations) | 1
Acute gastroenteritis (Gastrointestinal disorders) | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Worsening arrhythmia (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Worsening coronary artery disease (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1 — Led to shortness of breath and altered mental status.
Blocked fistula (Vascular disorders) | 1
Flu (Infections and infestations) | 1
Blocked artery (Vascular disorders) | 1
Accelerated hypertension (Vascular disorders) | 1
Osteomyelitis (Infections and infestations) | 1 — Caused by a MRSA infection.
Depression (Psychiatric disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRN (Pro re Nata) (N=60)
Vitreous hemorrhage (Eye disorders) | 9
Neovascularization elsewhere (Eye disorders) | 2
Neovascularization of the disc (Eye disorders) | 1
Worsening cataract (Eye disorders) | 8
Corneal abrasion (Eye disorders) | 1
Subconjunctival hemorrhage (Eye disorders) | 1
Superficial punctate keratitis (Eye disorders) | 1
Eye swelling post-cataract extraction (Eye disorders) | 1
Posterior vitreous detachment (Eye disorders) | 1
Floaters (Eye disorders) | 5
Visual disturbance (Eye disorders) | 1
Epiphora (Eye disorders) | 1
Posterior capsule opafication (Eye disorders) | 1
Iritis (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Vitreous debris (Eye disorders) | 1
Optic nerve pallor (Eye disorders) | 1
Decreased vision (Eye disorders) | 4
Ocular sensitivity (Eye disorders) | 5

LIMITATIONS AND CAVEATS:
Limitations of the ENDURANCE study include the small population and employment of aflibercept re-treatment criteria that allowed physicians to use their varying clinical judgement in determining anti-VEGF re-treatment instead of a strict protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No